CLINICAL TRIAL: NCT02266121
Title: Improving Cognitive Aptitudes With tDCS in Patients With Multiple Sclerosis / Améliorer Les capacités Cognitives Par tDCS Chez Les Patients Souffrants de sclérose en Plaques
Brief Title: Improving Cognitive Aptitudes With tDCS in Patients With Multiple Sclerosis
Acronym: MScog-tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitement
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Université Catholique de Louvain (Other); Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B039201421534
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Secondary-progressive Multiple Sclerosis; Cognitive Deficits; Motor Deficits
Keywords: Multiple Sclerosis; MS; Cognitive deficits; Motor deficits; Fatigue; Nervous System Diseases; Brain Diseases; Brain stimulation; Working memory; Motor learning; Central Nervous System Diseases; Neuropsychological rehabilitation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Cognition Disorders; Neurologic Manifestations; Multiple Sclerosis; Fatigue; Nervous System Diseases; Brain Diseases; Central Nervous System Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- real tDCS (Active Comparator): Patients will receive non-invasive and painless brain stimulation over the rain areas involved in cognitive aptitudes.
  tDCS will be applied during 20 minutes while patients will perform attentional, working memory and executive tasks
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): this will be exactly as for "real tDCS" unless that the tDCS will be rapidly turned off, unbeknown from patients-therapist-examinator (double-blind trial)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Device: transcranial direct current stimulation tDCS tdcs (ELDITH, Neuroconn, Ilmenau, Germany)

SUMMARY:
Noninvasive brain stimulations (NIBS) will be used in MS patients with cognitive impairments to enhance their cognitive aptitudes.

DETAILED DESCRIPTION:
tDCS will be used in a sham-controlled, double-blind, randomized, cross-over control trial in MS patients suffering from cognitive impairments and/or motor deficits. After informed consent and recruitment, patients will be randomly (computer method) allocated to real or sham tDCS, that will be applied during working memory and attentional tasks. A few days/weeks after completing one arm, the patients will enter the other arm (double-blind cross-over design).

Baseline and follow-up outcomes about cognitive aptitudes, motor tasks and fatigue will be collected.

ELIGIBILITY:
Inclusion Criteria:

* MS patients with relapsing remitting MS/secondary progression MS (based on the 2010 revised McDonald criteria)
* Cognitive deficits
* Motor deficits

Exclusion Criteria:

* contraindication to tDCS (seizure or epilepsy, metal in the head, …)
* major psychiatric conditions or major depression
* coexisting instable medical condition
* substance or alcohol abuse
* regular intake of drug that strongly modulate brain excitability
* major sequels from MS preventing participation in the study
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Enhancement of Cognitive aptitudes with tDCS | from baseline to 4 weeks after the intervention
  The effect of intervention on attentional, working memory and executive function deficits will be quantified by means of validated tests before and after intervention.

SECONDARY OUTCOMES:
Enhancement of Motor skills with tDCS | from baseline to 4 weeks after the intervention
  Performance on motor skill learning tasks and on different commonly used tasks (Purdue Pegboard, hand dynamometer, pinch dynamometer, 9-HPT, motor skill learning with a videogame, ...) will be measured to explore the impact of tDCS on these parameters in MS patients' population.
Impact on Fatigue and Enhancement of Cognitive performances with tDCS | from baseline to 4 weeks after the intervention
  The effect of intervention on fatigue and performances on the cognitive tasks will be quantified by means of validated questionnaires at inclusion and after tDCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, CHU Dinant Godinne UcL Namur, Yvoir, Namur, Belgium